CLINICAL TRIAL: NCT01404767
Title: Tight Hemodynamic Control in Patients Who Are Chronically on Metoprolol: A Study Comparing the Post Op Continuation of the Preoperative Oral Dose Beta Blockers to Intravenous Esmolol Titrated to a Target Heart Rate (HR)
Brief Title: Tight Hemodynamic Control in Patients Who Are Chronically on Metoprolol
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment slow over 2 years a change in the population less on metoprolol than initially anticipated
Sponsor: University Health Network, Toronto (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-0713-A
Record Dates: First submitted 2011-06-21; First posted 2011-07-28 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Vascular Disease; Hypertension; Angina; Cardiac Disease
Keywords: Vascular surgery; esmolol; hemodynamic control
MeSH Terms: conditions — Vascular Diseases; Hypertension; Angina Pectoris; Heart Diseases | interventions — esmolol; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metoprolol oral dose or Placebo infusion (Active Comparator)
  Interventions: Drug: Metoprolol
- Esmolol infusion or Placebo oral dose (Experimental)
  Interventions: Drug: Esmolol

INTERVENTIONS:
Drug: Esmolol — Baseline treatment consists of a bolus of 500ug/kg/min followed by an infusion of 50ug/kg/min for 4 minutes and titrating in increment of 50ug/kg/min up to a maximum of 300ug/kg/min to maintain a HR within 10% of the target HR (≤ 70 bpm), which is 70± 7 bpm.
  Arms: Esmolol infusion or Placebo oral dose
Drug: Metoprolol — The night and morning before surgery, the patients in the metoprolol arm will receive their standard dose of beta blocker metoprolol.These patients will receive their daily beta blockers orally or via nasogastric tube postoperatively if they are NPO (Group A).
  Arms: Metoprolol oral dose or Placebo infusion

SUMMARY:
This study proposes to assess the effect of the standard of care, which is continuation of the pre op beta blocker dose into the post operative period compared to the administration of esmolol titrated to a pre determined target HR. The primary outcome will compare postoperative plasma levels of metoprolol in 2 cohorts in a group who has been continued on metoprolol (administrated via a nasogastric tube in NPO patients) to a group who has been withdrawn from metoprolol but given an esmolol infusion titrated to HR. Secondary outcomes will compare a) the hemodynamic responses, documenting the incidence of unplanned hypotension and bradycardia and b) to compare the effects of Heart rate to the incidence of myocardial ischemia, arrhythmias, delirium and infarction.

DETAILED DESCRIPTION:
The number of high-risk patients undergoing non-cardiac surgery has increased continuously over the last two decades. There is a paucity of data exist about the bioavailability of postoperative administrated beta-blockers. One study reported adequate plasma levels of Propanolol after administration via nasogastric tube but not after oral administration in patient undergoing thyroid surgery.Thus it is possible that patients maintained on oral beta blockers may in fact be experiencing a withdrawal syndrome. Because of the importance of avoiding withdrawal of beta blockers, intravenous administration may be the only alternative in cases where oral administration fails to achieve adequate plasma levels perioperatively. Furthermore, due to changes in pharmacodynamics, intravenous dosage may be the optimal way to achieve tight hemodynamic control. There is, however, no data on the post-operative hemodynamic effects of orally administered beta blockers in patients on chronic beta blockers.

ELIGIBILITY:
Patient inclusion criteria:

* Elective vascular surgery
* Any of the following co morbidities

  * Diabetes
  * Angina
  * Congestive heart failure
  * A serum creatinine above 176 mmol/l
* All patients must be on stable dose of oral metoprolol (≥ 30 days)
* Age ≥ 20 years and ≤ 80 years
* Written informed consent to participate to the study

Patient exclusion criteria:

* Inability to understand the study protocol
* Prior gastric surgery or small bowel resection
* Pacemaker ( since it precludes the measurement of ST changes)
* Malabsorption syndromes
* Body Mass Index < 18 and > 35
* Any patient with suspected of diagnosed Cerebral vascular disease. (We chose to exclude CVA patients due to the ongoing controversy about the increased incidence of stroke in patients have surgery and who are taking beta-blockers.)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-04; Primary Completion 2011-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The difference between plasma levels of metoprolol within two groups | 0,1, 2, 4, 8, 12, 24 hours post intervention
  Comparisons measured in the pre-operative to intra-operative and post operative periods within metoprolol arm as well as between esmolol arm and metoprolol arm. Plasma levels will be correlated with both the hemodynamic response (HR) and the incidence of postoperative ischemia. The covariates (HR, BP, HR variability, etc) on PK/PD correlation will be examined.

SECONDARY OUTCOMES:
The amount of time the target heart rate is maintained and the incidence of perioperative hypotension and bradycardia. | Data will be recorded for 48 hours from arrive to the recovery area
  Additional assessments include cardiovascular morbidity and mortality including 30-day mortality, myocardial infarction, new cardiac arrhythmia, congestive heart failure, and renal failure, the incidence of post operative delirium, transient ischemic attack, stroke, and length of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Beattie, MD, FRCP, Principal Investigator — University Health Network, Toronto General Hospital
Locations (1):
- University Heatlh Network, Toronto General Hopsital, Toronto, Ontario, Canada